CLINICAL TRIAL: NCT00759018
Title: Expanded Access of Prochymal (Ex-vivo Cultured Adult Human Mesenchymal Stem Cells) Infusion for the Treatment of Pediatric Patients Who Have Failed to Respond to Steroid Treatment for Acute GVHD
Brief Title: Prochymal Expanded Access Treatment for Pediatric Patients Who Have Failed Steroids for Acute GVHD
Status: No longer available | Type: Expanded Access
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Other Study IDs: 275
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Graft vs Host Disease; Graft-Versus-Host Disease
Keywords: GVHD; Prochymal; Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — remestemcel-l

INTERVENTIONS:
Biological: remestemcel-L — Patients will be treated with Prochymal® twice per week at a dose of 2 x 10^6 hMSC/kg (actual body weight) for each of 4 consecutive weeks. Infusions will be administered at least 3 days apart.
  Other Names: Prochymal®; Ex-vivo Cultured Adult Human Mesenchymal Stem Cells

SUMMARY:
This protocol allows for the treatment of pediatric patients, male and female, between the ages of 2 months and 17 years. Patients must have failed steroid treatment for Grade B-D acute GVHD.

DETAILED DESCRIPTION:
For the treatment of pediatric patients who have failed to respond to steroid treatment for acute graft-versus-host disease (GVHD). Failing steroid treatment for acute GVHD is defined as any Grade B-D (IBMTR grading) of acute GVHD that is not improving after at least 3 days of methylprednisolone (≥ 1 mg/kg/day) or equivalent.

Patients will be treated with Prochymal twice per week at a dose of 2 x 10^6 hematopoietic stem cells (hMSC)/kg (actual body weight) for each of 4 consecutive weeks. Infusions will be administered at least 3 days apart.

ELIGIBILITY:
Inclusion criteria:

* Patients must sign an informed consent form (ICF) before any protocol-related procedures, including any pre-treatment procedures, are performed.
* Since patients being treated with Prochymal® under this protocol are under 18, a parental signature of informed consent will be required.
* Patients must be 2 months to 17 years of age, inclusive.
* Patients must have failed to respond to steroid treatment for Grades B-D acute GVHD • Failure to respond to steroid treatment for acute GVHD is defined as any Grade B-D acute GVHD that is not improving after at least 3 days of methylprednisolone (≥1 milligram per kilogram per day [mg/kg/day]) or equivalent.

Exclusion criteria:

* Patient must not have a known allergy to bovine or porcine products.
* Patient must not have received a transplant for a solid tumor disease.
* Patients must not have evidence of a pulmonary infiltrate or diffuse alveolar hemorrhage and must be unlikely to require more than 2 liters (L) of oxygen via face mask or an estimated fraction of inspired oxygen (FiO2) of 28% via other delivery methods in order to sustain an O2 saturation of 92% during the next 3 days.

Ages: 2 Months to 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, Study Director — Mesoblast, Inc.
Locations (27):
- United States (24):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Orange County, Orange, California
  - UCSF, San Francisco, California
  - Children's National, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Childrens Memorial, Chicago, Illinois
  - James Witcomb Riley Hosptial for Children, Indianapolis, Indiana
  - LSU Health Science Center/Children's Hospital, New Orleans, Louisiana
  - Wayne State University/Childrens' Hospital, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Doernbecher Children's Hospital (OHSU), Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Childrens Hospital, Houston, Texas
  - Methodist Childrens Hospital of South Texas, San Antonio, Texas
  - Massey Cancer Center, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Kurtzberg J, Prockop S, Chaudhury S, Horn B, Nemecek E, Prasad V, Satwani P, Teira P, Hayes J, Burke E; MSB-275 Study Group. Study 275: Updated Expanded Access Program for Remestemcel-L in Steroid-Refractory Acute Graft-versus-Host Disease in Children. Biol Blood Marrow Transplant. 2020 May;26(5):855-864. doi: 10.1016/j.bbmt.2020.01.026. Epub 2020 Feb 7. PMID 32044400